CLINICAL TRIAL: NCT01574443
Title: Brain Dynamics in Different Stages of Arousal and Anesthesia
Acronym: ECOG
Status: Terminated | Type: Observational
Why Stopped: Feasibility issues for subject recruitment and PI left the institution
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1106011763
Record Dates: First submitted 2012-03-16; First posted 2012-04-10 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Epilepsy
Keywords: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- epilepsy resection patients: Patients undergoing resection for refractory epilepsy

SUMMARY:
The principle aim of this project is to characterize the changes in relative stability of the intrinsic brain dynamics during onset of sleep and induction of general anesthesia. The investigators hypothesize that brain dynamics in the awake state are critical akin to physical systems close to a second order phase transition and that during loss of consciousness the dynamics move away from the critical point.

DETAILED DESCRIPTION:
1. Once the electrode array is placed during the first surgery (on the day of admission) we will record brain activity as subjects are waking up from anesthesia
2. While subjects are staying at New York Presbyterian hospital before the second surgery we will record brain activity. Most of the recordings will be performed as subjects are going to sleep naturally, but other recordings will be acquired during waking hours. This will not interfere with normal monitoring of seizure activity.
3. Final recording session is immediately before the second operation as general anesthesia is gradually induced. During this time subjects may be asked to follow simple commands like: "Open your eyes" in order to determine the level of consciousness. Also during this session, if arterial line is placed by the anesthesiologist for real-time blood pressure monitoring we will collect several small (~1 ml) blood samples to determine blood concentration of anesthetics. Approximately 1 teaspoon of blood will be obtained in total. No additional venipuncture will be necessary.

No additional invasive procedures will be performed for the purposes of the study. We will use the same electrode array as is typically used for monitoring and mapping of epilepsy. Subjects will receive the same anesthetic agent as is commonly used for induction of anesthesia for this surgery (propofol). Subjects will be monitored in the same way as is normally done during surgical procedures and during your stay at New York Presbyterian hospital.

As a part of the study subjects may be asked simple questions as they go under anesthesia.

We may collect several small blood samples (described above) to determine the concentration of anesthetic agents.

ELIGIBILITY:
Inclusion Criteria:

1.Patients referred for epilepsy resection surgery with Dr. Theodore Schwartz

Exclusion Criteria:

1. Patient refusal.
2. Patients requiring rapid sequence induction because of concerns about delayed gastric emptying as a result of diabetes or other medical conditions.
3. Age less than 15 or greater than 65 years old.
4. Pregnant or nursing.
5. Inability to follow simple commands such as "Open your eyes" and "Squeeze my hand" for any reason.
6. Severe mental disability.
7. Allergy to propofol or any components of the formulation.
8. Poor suitability for propofol infusion because of other medical concerns such as severe heart disease.
9. Patients deemed to have a difficult airway thus necessitating awake fiberoptic intubation.
10. Patients with severe sleep apnea requiring CPAP/BiPAP.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing epilepsy resection surgery
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2011-08-22 (Actual); Primary Completion 2015-05-11 (Actual); Study Completion 2016-04-08 (Actual)

PRIMARY OUTCOMES:
Characterization of changes in brain dynamics during induction of anesthesia, using electrocorticography (ECoG). | < 1 hour
  The patterns of electrical activity during induction and emergence from anesthesia will be compared to what is recorded during natural sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Kane Pryor, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital/ Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No